CLINICAL TRIAL: NCT00753948
Title: The Effect of Nitric Oxide on Pulmonary Resistances and Blood Pressure in Persons With Tetraplegia
Brief Title: Exhaled Levels of Nitric Oxide
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B4335-V
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Tetraplegia; Asthma
Keywords: Tetraplegia; Mild asthma; Exhaled Nitric Oxide; NOS inhibitor; Spinal cord injury; Pulmonary Function
MeSH Terms: conditions — Quadriplegia; Asthma; Spinal Cord Injuries | interventions — NG-Nitroarginine Methyl Ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chronic Tetraplegia (Experimental): Individuals with chronic tetraplegia
  Interventions: Drug: N-Nitro L-arginine-methylester (L-NAME)
- Mild Asthma (Active Comparator): Individuals with diagnosed mild asthma
  Interventions: Drug: N-Nitro L-arginine-methylester (L-NAME)
- Healthy Control (Placebo Comparator): Neurologically intact, otherwise healthy, age-matched control
  Interventions: Drug: N-Nitro L-arginine-methylester (L-NAME)

INTERVENTIONS:
Drug: N-Nitro L-arginine-methylester (L-NAME) — A non-specific inhibitor of the nitric oxide synthase enzyme.

SUMMARY:
Previously it was observed that individuals with tetraplegia have reduced baseline airway caliber and exhibit non-specific airway hyperresponsiveness (AHR). In persons with tetraplegia we have suggested that this is due to overriding cholinergic airway tone. In asthma, the mechanisms underlying bronchoconstriction and AHR are more closely tied to airway inflammation. Whether AHR in tetraplegia is also related to chronic airway inflammation is unknown.

Recently, a non-invasive technique for assessing airway inflammation has been established in asthma that involves measurement of nitric oxide (NO) concentrations (FeNO) in expired air. FeNO is elevated in asthma likely due to excess NO production by inflammatory cells within the airway Measurement of FeNO in persons with tetraplegia would help in assessing the role of airway inflammation in this population. This may have therapeutic significance in such individuals. NO in the lung is felt to be the principal inhibitory neurotransmitter of the non-adrenergic, non-cholinergic (NANC) system. It is thought that inhalation of NO has no effect on airway tone in healthy individuals but reduces methacholine responsiveness while having weak direct bronchodilatory effect in asthmatics.

The primary purpose of this study is to determine the levels of exhaled NO (FeNO) in individuals with chronic cervical spinal cord injury (SCI), and to compare them with those obtained in age and sex matched able-bodied individuals and subjects with stable mild to moderate asthma. If the FeNO levels are high and comparable to those found in asthmatic subjects, this will imply the role of chronic inflammation in reduced baseline airway caliber and non-specific airway hyper-responsiveness (AHR) exhibited by individuals with chronic cervical SCI. If the FeNO levels are comparable with those found in able-bodied controls, this will support our previous statement that unopposed cholinergic innervation is responsible for low baseline airway caliber and AHR in individuals with chronic tetraplegia. Further scientific conclusions about NO and its role in control of airway tone, pulmonary resistances and blood pressure will be drawn upon intravenous and inhaled administration of L-NAME. This compound has been shown promising results for the treatment and prevention of orthostatic hypotension in individuals with tetraplegia. Knowing its effects on airways and potential of easier mode of delivery (inhalation vs. intravenous) is of utmost importance.

DETAILED DESCRIPTION:
The study requires a maximum of five study visits in the following order: 1. nebulized normal saline, 2. nebulized 1mg/kg of L-NAME (see below), 3. intravenous normal saline, 4. intravenous 1 mg/kg L-NAME, 5. intravenous 2 mg/kg L-Name.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Age between 18 and 65 years.
3. Able-bodied individuals, persons with mild asthma or individuals with tetraplegia for at least one year of duration.
4. Able to perform acceptable pulmonary function tests and follow procedures.

Exclusion Criteria:

1. coronary artery disease;
2. active cigarette smokers or previous smokers who stopped <5 years ago;
3. MI or stroke within 3 months;
4. moderate to severe reduction in lung function defined as FEV1 < 70 % predicted (except in individuals with tetraplegia);
5. hypertension;
6. medications known to affect the cardiovascular system;
7. pregnancy
8. current use of cholinesterase medication; and
9. lack of mental capacity to give informed consent Group specific exclusion criteria for

Asthmatic subjects:

1. Moderate to severe disease as per spirometric indices;
2. testing within 48 hours of last administration of long acting inhaled bronchodilator;
3. testing within 7 days of last administration of glucocorticoids;
4. testing within > 24 hours since last administration of leukotriene modifiers; and
5. testing within 8 hours of last administration of a short acting bronchodilator medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Radulovic, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Radulovic M, Schilero GJ, Wecht JM, La Fountaine M, Rosado-Rivera D, Bauman WA. Exhaled nitric oxide levels are elevated in persons with tetraplegia and comparable to that in mild asthmatics. Lung. 2010 Jun;188(3):259-62. doi: 10.1007/s00408-009-9207-x. Epub 2009 Dec 15. PMID 20012982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from SCI service of James J. Peters VAMC as well as from SCI outpatient clinics. Participants in the asthma group were recruited through medicine clinic at James J. Peters VAMC. Healthy able-bodied controls were recruited from the group of able-bodied controls that has been doing studies with our center in the past.
Groups:
- Chronic Tetraplegia: Individuals with chronic tetraplegia
  N-Nitro L-arginine-methylester (L-NAME) : A non-specific inhibitor of the nitric oxide synthase enzyme.
- Mild Asthma: Individuals with diagnosed mild asthma
  N-Nitro L-arginine-methylester (L-NAME) : A non-specific inhibitor of the nitric oxide synthase enzyme.
- Healthy Control: Neurologically intact, otherwise healthy, age-matched control
  N-Nitro L-arginine-methylester (L-NAME) : A non-specific inhibitor of the nitric oxide synthase enzyme.
Period: Overall Study
Arm/Group | Chronic Tetraplegia | Mild Asthma | Healthy Control
Started | 9 | 7 | 7
Completed | 9 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Controls: Neurologically intact, otherwise healthy, age-matched control
  N-Nitro L-arginine-methylester (L-NAME) : A non-specific inhibitor of the nitric oxide synthase enzyme.
- Total: Total of all reporting groups
Arm/Group | Chronic Tetraplegia | Mild Asthma | Healthy Controls | Total
Number analyzed (Participants) | 9 | 7 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 7 | 7 | 23
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (10) | 42 (9) | 37 (10) | 40 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 8 | 6 | 6 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 7 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Exhaled Levels of Nitric Oxide
Description: Nitric Oxide was measured applying a real time technique for measurement of Nitric Oxide in Exhaled Breath Condensate. Elevated Nitric Oxide in exhalate is a measure of elevated production of NO in conditions such as underlying inflammation and/or oxidative stress. Exhaled NO was reported as the mean of three values within 10% of each other.
Time Frame: Exhaled NO reported during visit, before intervention at baseline, post intervention at 60 minutes and 120 minutes
Measure: Mean (Standard Deviation); unit: ppb (parts per bilion)
Arm/Group | Chronic Tetraplegia | Mild Asthma | Healthy Controls
Number analyzed (Participants) | 7 | 3 | 7
ppb (parts per bilion)
  Baseline (before intervention) | 17.27 (4.96) | 19.83 (8.15) | 15.025 (9.75)
  60 minutes (post intervention) | 3.70 (3.14) | 5.56 (2.93) | 4.07 (3.47)
  120 minutes (post intervention) | 3.04 (2.23) | 5.73 (3.70) | 3.71 (3.46)

2. Secondary Outcome: Specific Airway Conductance (sGaw) as Measured by Plethysmography
Description: Specific airway conductance (sGaw) is the airway conductance relative to lung volume because it takes into account the important effect of lung volume on airway resistance, it is a useful index of bronchomotor tone.
Time Frame: Specific airway conductance reported during visit, before intervention at baseline, post intervention at 60 minutes and 120 minutes
Measure: Mean (Standard Deviation); unit: L/sec/cmH20/L
Arm/Group | Chronic Tetraplegia | Mild Asthma | Healthy Controls
Number analyzed (Participants) | 7 | 1 | 7
L/sec/cmH20/L
  Baseline (before intervention) | 0.164 (0.071) | 0.336 (0) | 0.197 (0.043)
  60 minutes (post intervention) | 0.218 (0.093) | 0.315 (0) | 0.196 (0.047)
  120 minutes (post intervention) | 0.207 (0.094) | 0.345 (0) | 0.197 (0.043)

ADVERSE EVENTS:
Arm/Group | Chronic Tetraplegia | Mild Asthma | Healthy Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes